CLINICAL TRIAL: NCT06309186
Title: Empowerment and Burnout of Midwives at the End of Health Emergency From SARS-CoV2: a Cross-sectional Observational Study in Friuli-Venezia Giulia Region
Brief Title: Empowerment and Burnout of Midwives at the End of Health Emergency From COVID-19
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 30/2023
Record Dates: First submitted 2024-03-12; First posted 2024-03-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: COVID-19
Keywords: Midwifery; Empowerment; Burnout
MeSH Terms: conditions — COVID-19; Empowerment; Burnout, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Midwives: The study involves a convenience sample of midwives registered with the two Orders of the Midwifery Profession in Friuli-Venezia Giulia Region (Italy)
  Interventions: Other: Evaluation of midwifes' burnout

INTERVENTIONS:
Other: Evaluation of midwifes' burnout — Burnout evaluated by questionnaires

SUMMARY:
As the fifth wave of COVID-19 comes to an end and the pandemic's countermeasures expire, there is a need to assess the impact of the pandemic on health care providers, especially midwives, as the professionals deputed to promote and protect women's holistic health, in all phases, physiological and otherwise, of the life cycle. The midwife considers the person as a whole, in which the mind-body-culture components interact profoundly. Prevention and containment measures have impacted on midwifery clinical and nursing practices with the mandatory continuous use of personal protective equipments (PPE) and social distancing to protect the patient and the practitioner, effectively hindering the intimacy of the woman-midwife relationship. The impact assessment focuses on two dimensions: learning, investigated as perceived empowerment, and perceived malaise, investigated as burnout. Empowerment has a positive connotation, which can offset burnout, a syndrome that affects the physical, psychological and emotional health of midwives and can have significant negative implications on midwife turnover, patient safety and outcomes, and the efficiency of healthcare organisations.

ELIGIBILITY:
Inclusion Criteria:

1. Midwives registered in the orders of Friuli Venezia Giulia (FVG) region
2. Midwives in practice for at least one year
3. Midwives practicing in FVG region

Exclusion Criteria:

1. Consent not granted
2. Midwives in retirement for more than a year

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Midwives
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of empowerment of midwives | At enrolment
  Midwives empowerment will be evaluated with the italian validated version of the "Perceptions of empowerment in midwifery scale-revised" (PEMSR). It consists of 19 items, expressing 4 subscales divided into four subscales: autonomy/empowerment (4 items); manager support (5 items); professional recognition (5 items); and skills and resources (5 items). Total scores are calculated for each of the subscales by summing all the scores from each item, and then dividing by the number of items in the same subscale. Scores range from 1 (low level of empowerment), to 5 (high level of empowerment).
Number of midwives affected by burnout | At enrolment
  Burnout will be evaluated with the Maslach Burnout Inventory (MBI), an instrument of 22 Likert items of 7 points on feelings related to work. Respondents rate how often they experience these feelings on a 7-point Likert scale from 0 (never) to 6 (every day). The MBI includes 3 subscales or dimensions: emotional exhaustion (EE), depersonalization (DP, and personal accomplishment (PA). Higher item scores in EE and DP and low in PA correspond to high levels of burnout.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste
  - Ordine delle ostrtriche di Trieste e Gorizia, Trieste

IPD SHARING:
Plan to Share IPD: Undecided